CLINICAL TRIAL: NCT05668611
Title: Design and Evaluation of a Train the Trainer Curriculum to Scale Up Automated Intelligence Supported Echocardiography for Rheumatic Heart Disease Screening in a Public Health Care System
Brief Title: Train the Trainer Curriculum to Scale up AI Supported Echo for RHD Screening in a Public Health System
Acronym: ADD-RHD 2B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Uganda Heart Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-0312
Record Dates: First submitted 2022-10-26; First posted 2022-12-30 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Rheumatic Heart Disease
MeSH Terms: conditions — Rheumatic Heart Disease

STUDY DESIGN:
Intervention Model Description: This is a two-phase cohort study that will determine the ability of MOH nurses to accurately integrate echocardiographic screening for rheumatic heart disease into primary healthcare clinics in Uganda.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Training (Experimental): 4 Ministry of Health nurses will be trained by expert trainers to become certified in focused echocardiography acquisition and interpretation in order to screen patients for rheumatic heart diseases
  Interventions: Other: Primary Training Phase; Other: Primary Assessment Phase; Other: Primary Screening Phase
- Secondary Training (Experimental): The 4 Ministry of Health nurses trained in Aim 1 will then train and certify 3 other nurses from their clinics in focused echocardiography acquisition interpretation.
  Interventions: Other: Secondary Training Phase; Other: Secondary Assessment Phase; Other: Secondary Screening Phase

INTERVENTIONS:
Other: Primary Training Phase — A four-day training program taken over the course of two weekends will include materials on RHD and RHD echocardiographic screening using focused artificial intelligence navigational guided echocardiographic acquisition to identify patients who are screen positive or screen negative for RHD. The echo protocol will be limited to the parasternal long axis-view (2D and color Doppler) focusing on mitral and aortic valve morphology and function and a single 2D apical 4 chamber view for auto EF. The curriculum package will include online modules, instructor delivered PowerPoint presentations, and hands on practice on volunteers with and without RHD.
  Arms: Primary Training
Other: Primary Assessment Phase — A pre- and post-training test on RHD knowledge and diagnosis will be administered. A rapid competency assessment, including obtaining imaging on volunteers with or without RHD and an online test with pre-recorded cases of RHD, LV dysfunction and Pericardial effusions, will be utilized at the end of the 4-day training sessions. Trainees will be monitored by trained study personnel and at the end of the practicum training, the expert users will blindly review and assess the quality of each study using the standardized scale and competency scorecard provided below. Additionally, they will be asked to pass the knowledge quiz (80% or better). If competency is not achieved, an additional weekend of training can be added.
  Arms: Primary Training
Other: Primary Screening Phase — Following certification, the certified MOH nurses will integrate echocardiographic screening into the routine workflow at the 4 HCIII/IV clinics with each nurse carrying out screening at the assigned HC on patients (aged 5-40) presenting to the health center for routine care.
  Screening will be done daily over a period of one month. A minimum total of 400 participants will be screened during this period; each nurse will screen as many patients as they can, with a minimum of 100 participants (at least 5 participants per day). At the end of each screen, the trainees will interpret the screen as screen negative or screen positive. They will go ahead to refer participants identified as screen positives to the district hospital (LRRH) for a confirmatory echo.
  At the end of each screening day, all images will be uploaded to a cloud server for a confirmatory review by a cardiology fellow or cardiology attending physician, within in 1 - 2 weeks.
  Arms: Primary Training
Other: Secondary Training Phase — Each Primary Trained MOH Nurse will train 3 other nurses from their Health Center using pre-recorded PowerPoints.
  Arms: Secondary Training
Other: Secondary Assessment Phase — The secondarily trained nurses will be assessed and certified by the nurse trainer.
  Arms: Secondary Training
Other: Secondary Screening Phase — Following certification, the certified MOH nurses will integrate echocardiographic screening into the routine workflow at the 4 HCIII/IV clinics with each nurse carrying out screening at the assigned HC on patients (aged 5-40) presenting to the health center for routine care.
  Screening will be done daily over a period of two months. A minimum total of 1200 participants will be screened during this period; each nurse will screen as many patients as they can, with a minimum of 100 participants. At the end of each screen, the trainees will interpret the study as screen negative or screen positive. They will go ahead to refer participants identified as screen positives to the district hospital (LRRH) for a confirmatory echo.
  At the end of each screening day, all images will be uploaded to a cloud server for a confirmatory review by a cardiology fellow or cardiology attending physician, within in 1 - 2 weeks.
  Arms: Secondary Training

SUMMARY:
The first primary objective of this study is to determine the diagnostic performance (sensitivity and specificity) of primary MOH nurses who have completed certification in focused echocardiography acquisition and interpretation by expert trainers to accurately identify patients who are screen positive and screen negative for rheumatic heart disease. The second primary objective is to determine the diagnostic performance (sensitivity and specificity) of secondary MOH nurses who have completed certification in focused echocardiography acquisition and interpretation by MOH nurse trainers to accurately identify patients who are screen positive and screen negative for rheumatic heart disease.

DETAILED DESCRIPTION:
Objective 1:

4 ultrasound naïve nurses (Primary) employed at the HCIII/IVs participating in ADD-RHD Part 1 (SOMREC REF 2021-61) in Lira, will be trained and certified by experts in echocardiography for RHD on focused RHD echocardiographic screening examination and interpretation using a novel AI guided software.

Focused RHD screening echocardiograms by the 4 nurses will be integrated into routine clinical practice at their assigned HCIII/IVs for 1 month.

Screen positive patients will be referred to LRRH for confirmatory echocardiogram using a Standard echocardiographic machine under the National RHD registry (SOMREC REF 2014-137).

All echocardiograms will be uploaded to a secure cloud-based server and over-read by a cardiologist with in one - two (1 - 2) weeks to ensure patient safety and to determine trainee performance.

Diagnostic accuracy, sensitivity, specificity, positive and negative predictive values will be calculated.

4 MOH trainees will use pre-recorded PowerPoint presentations to conduct hands-on training for phase 2 (secondary) nurses.

Objective 2:

Similar to Phase 1 with just a few exceptions. 12 MOH nurses will be trained and certified by MOH nurse trainers from phase 1 to acquire and interpret RHD focused screening echocardiograms using a novel AI guided software.

Screening will be integrated into routine care for 2 months and diagnostic performance assessed.

ELIGIBILITY:
Inclusion Criteria:

* Attend same HCIII/IV sites that the MOH nurses work at
* Agree to participate via the study's informed consent

Exclusion Criteria:

* Very sick participants requiring transfer to higher level facility or inpatient care

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1628 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
RHD Echocardiographic Diagnostic accuracy, sensitivity, specificity of MOH nurses | 2 months after completion of training
  Diagnostic performance of MOH nurses who have completed certification in focused echocardiography acquisition and interpretation by expert trainers will be assessed. Diagnostic accuracy, sensitivity, specificity, positive and negative predictive values will be calculated to determine diagnostic performance of MOH nurses who have completed certification on focused echocardiography acquisition and interpretation. The ability of trainees to correctly identify screen positive and negative patients for RHD using known expert diagnosis as the reference. Correct determination of RHD screen positive/negative in at least 80% of cases is the benchmark

SECONDARY OUTCOMES:
Knowledge Assessment | Immediately before the training session and immediately after completion of training
  Questionnaire to test compare pre and post training knowledge about Rheumatic Heart Disease administered to nurse trainees.
Computer Based Testing | Immediately following training
  Computer based testing designed to determine positive and negative screening referrals of patients with RHD and other cardiac diseases
Rapid Competency assessment | Immediately following training
  This assessment will be administered post training to nurse trainees. It is an observation- based assessment designed to assess correct use of the technology, basic image acquisition proficiency, diagnostic accuracy and image quality.
Provider satisfaction | Immediately post training
  Surveys questions on training and screening experience along with guided discussions on the training and screening experiences will be administered to nurse trainees
Longitudinal Image Quality | Daily assessment for 1 month
  Expert Echocardiographers will access each image acquired by nurses using the ACEP scale. A scale of 1-5 (1) being no recognizable structure and (5) being excellent image quality of all structures. A score of 3 and above will be considered diagnostic.
Provider confidence | Daily assessment for 1 month
  Nurses will subjectively report their level of confidence regarding image quality. The levels of confidence will be assessed. (1) Very confident, image quality is good and adequate for diagnosis. (2) Fairly confident, image is good but confirmation of diagnosis by expert trainer needed, (3) Not confident, image quality not adequate.
Diagnostic performance for other common categories of cardiac diseases | Through completion of screening phase, average of 1 month
  Assess nurse's ability to accurately identify left ventricular dysfunction and pericardial effusion as compared to the same standard applied by an expert.
Time to certification | Trough first day of training to study completion, average of 1 year
  Determine the time from the first day of training to certification for participants including remediation time.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Z Beaton, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Uganda Heart Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No